CLINICAL TRIAL: NCT06173557
Title: Intraoperative Measurement Technique for Improved Accuracy of Femoral Offset and Leg Length in Total Hip Replacement: A Retrospective Cohort Study
Brief Title: Intraoperative Measurement Technique
Acronym: THR
Status: Completed | Type: Observational
Sponsor: Ziv Medical Center (Other)
Responsible Party: Principal Investigator, David Rothem, Head of orthopedic department, Ziv Medical Center
Other Study IDs: ZivMC; 0025-15-ziv (Registry Identifier: ZivMC)
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Total Hip; Limb Length Discrepancy
Keywords: total hip replacement; limb length discrepancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: entailed calculation of the distances between reference points on the ischium, greater trochanter, and the screwdriver. Measurements were collected from radiographic i — technique of intraoperative measurement of the femoral offset and limb length was used, entailed calculation of the distances between reference points on the ischium, greater trochanter, and the screwdriver. Measurements were collected from radiographic imaging data and surgical reports

SUMMARY:
This retrospective cohort study included 50 consecutive patients who underwent THR. All surgeries were performed by the same orthopedic surgeon, using posterior approach. In all patients, the same technique of intraoperative measurement of the femoral offset and limb length was used, entailed calculation of the distances between reference points on the ischium, greater trochanter, and the screwdriver. Measurements were collected from radiographic imaging data and surgical reports.

DETAILED DESCRIPTION:
Introduction: Restoration of limb length equality and femoral offset is critical for the success of THR. The purpose of this study was to investigate the efficacy of a novel intraoperative measurement technique in minimizing errors in leg length and offset in total hip replacement (THR).

Methods: This retrospective cohort study included 50 consecutive patients who underwent THR. All surgeries were performed by the same orthopedic surgeon, using posterior approach. In all patients, the same technique of intraoperative measurement of the femoral offset and limb length was used, entailed calculation of the distances between reference points on the ischium, greater trochanter, and the screwdriver. Measurements were collected from radiographic imaging data and surgical reports.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent THR due to primary osteoarthritis of the hip joint.

Exclusion Criteria:

* Patients who underwent THR for any other reasons
* patients that underwent revision surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50 consecutive patients who were admitted to the orthopedic department for elective THR
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
outcome | 1 year
  calculation of the distances between reference points on the ischium, greater trochanter, and the screwdriver

IPD SHARING:
Plan to Share IPD: No
no sharing